CLINICAL TRIAL: NCT02872116
Title: A Randomized, Multicenter, Open-Label, Phase 3 Study of Nivolumab Plus Ipilimumab or Nivolumab in Combination With Oxaliplatin Plus Fluoropyrimidine Versus Oxaliplatin Plus Fluoropyrimidine in Subjects With Previously Untreated Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer
Brief Title: Efficacy Study of Nivolumab Plus Ipilimumab or Nivolumab Plus Chemotherapy Against Chemotherapy in Stomach Cancer or Stomach/Esophagus Junction Cancer
Acronym: CheckMate649
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-649; 2016-001018-76 (EudraCT Number)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer; Esophageal Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Nivolumab; Ipilimumab; Oxaliplatin; Capecitabine; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nivolumab + Ipilimumab (Experimental): Nivolumab + Ipilimumab for 4 doses, followed by Nivolumab monotherapy
  Enrollment is closed for this arm
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- XELOX (Oxaliplatin + Capecitabine) (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- FOLFOX (Oxaliplatin + Leucovorin + Fluorouracil) (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- Nivolumab + XELOX (Experimental)
  Interventions: Drug: Nivolumab; Drug: Oxaliplatin; Drug: Capecitabine
- Nivolumab + FOLFOX (Experimental)
  Interventions: Drug: Nivolumab; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Nivolumab + FOLFOX; Nivolumab + Ipilimumab; Nivolumab + XELOX
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Nivolumab + Ipilimumab
Drug: Oxaliplatin — Specified dose on specified days
  Arms: FOLFOX (Oxaliplatin + Leucovorin + Fluorouracil); Nivolumab + FOLFOX; Nivolumab + XELOX; XELOX (Oxaliplatin + Capecitabine)
Drug: Capecitabine — Specified dose on specified days
  Arms: Nivolumab + XELOX; XELOX (Oxaliplatin + Capecitabine)
Drug: Leucovorin — Specified dose on specified days
  Arms: FOLFOX (Oxaliplatin + Leucovorin + Fluorouracil); Nivolumab + FOLFOX
Drug: Fluorouracil — Specified dose on specified days
  Arms: FOLFOX (Oxaliplatin + Leucovorin + Fluorouracil); Nivolumab + FOLFOX

SUMMARY:
The main purpose of this study is to compare how long patients with gastric or gastroesophageal junction cancer live after receiving nivolumab and ipilimumab or nivolumab and chemotherapy compared with patients receiving chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Must have gastric cancer or gastroesophageal junction cancer that cannot be operated on and that is advanced or has spread out
* Did not receive neoadjuvant or adjuvant treatment (chemotherapy, radiotherapy, or both) for their disease within the last 6 months
* Must have full activity or, if limited, must be able to walk and carry out light activities such as light house work or office work
* Must agree to provide tumor tissue sample, either from a previous surgery or biopsy within 6 months or fresh, prior to the start of treatment in this study

Exclusion Criteria:

* Presence of tumor cells in the brain or spinal cord that have not been treated
* Active known or suspected autoimmune disease
* Any serious or uncontrolled medical disorder or active infection
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Any positive test result for hepatitis B or C indicating acute or chronic infection

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2031 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (179):
- United States (27):
  - Local Institution - 0005, Los Angeles, California
  - Local Institution - 0001, San Francisco, California
  - Local Institution - 0066, Aurora, Colorado
  - Local Institution - 0151, Denver, Colorado
  - Local Institution - 0136, Washington D.C., District of Columbia
  - Florida Cancer Specialists S., Fort Myers, Florida
  - Local Institution - 0147, Miami, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Local Institution - 0179, Marietta, Georgia
  - Local Institution - 0219, Arlington Heights, Illinois
  - Local Institution - 0120, Chicago, Illinois
  - Local Institution - 0021, Baltimore, Maryland
  - Local Institution - 0002, Boston, Massachusetts
  - Local Institution - 0135, Boston, Massachusetts
  - Local Institution - 0003, New York, New York
  - Local Institution - 0138, Cleveland, Ohio
  - Local Institution - 0186, Cleveland, Ohio
  - Local Institution - 0146, Eugene, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Local Institution - 0065, Pittsburgh, Pennsylvania
  - Local Institution - 0104, Nashville, Tennessee
  - Local Institution - 0140, Bedford, Texas
  - Local Institution - 0143, Dallas, Texas
  - Local Institution - 0213, Dallas, Texas
  - Local Institution - 0004, Houston, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Local Institution - 0150, Newport News, Virginia
- Argentina (7):
  - Local Institution - 0030, Caba, Buenos Aires
  - Local Institution - 0028, Capital Federal, Buenos Aires
  - Local Institution - 0029, Capital Federal, Buenos Aires
  - Local Institution - 0026, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0027, Córdoba
  - Local Institution - 0184, La Rioja
  - Local Institution - 0183, Viedma
- Australia (8):
  - Local Institution - 0202, Blacktown, New South Wales
  - Local Institution - 0100, Gosford, New South Wales
  - Local Institution - 0190, Southport, Queensland
  - Local Institution - 0101, Adelaide, South Australia
  - Local Institution - 0103, Ballarat, Victoria
  - Local Institution - 0102, Shepparton, Victoria
  - Local Institution - 0214, St Albans, Victoria
  - Local Institution - 0099, Perth, Western Australia
- Brazil (5):
  - Local Institution - 0053, Salvador, Estado de Bahia
  - Local Institution - 0046, Ijuí, Rio Grande do Sul
  - Local Institution - 0047, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0048, Barretos, São Paulo
  - Local Institution - 0054, São Paulo
- Canada (8):
  - Local Institution - 0035, Edmonton, Alberta
  - Local Institution - 0036, London, Ontario
  - Local Institution - 0067, Toronto, Ontario
  - Local Institution - 0052, Montreal, Quebec
  - Local Institution - 0196, Montreal, Quebec
  - Local Institution - 0051, Québec, Quebec
  - Local Institution - 0068, Sherbrooke, Quebec
  - Local Institution - 0034, Trois-Rivières, Quebec
- Chile (5):
  - Local Institution - 0032, Temuco, Región de la Araucanía
  - Local Institution - 0033, Viña del Mar, Región de Valparaíso
  - Local Institution - 0058, Independencia, Santiago Metropolitan
  - Local Institution - 0057, Santiago, Santiago Metropolitan
  - Local Institution - 0031, Santiago, Santiago Metropolitan
- China (22):
  - Local Institution - 0176, Beijing, Beijing Municipality
  - Local Institution - 0178, Beijing, Beijing Municipality
  - Local Institution - 0171, Beijing, Beijing Municipality
  - Local Institution - 0185, Fuzhou, Fujian
  - Local Institution - 0166, Guangzhou, Guangdong
  - Local Institution - 0160, Harbin, Heilongjiang
  - Local Institution - 0159, Zhengzhou, Henan
  - Local Institution - 0173, Changsha, Hunan
  - Local Institution - 0158, Changzhou, Jiangsu
  - Local Institution - 0154, Nanjing, Jiangsu
  - Local Institution - 0187, Nanjing, Jiangsu
  - Local Institution - 0156, Changchun, Jilin
  - Local Institution - 0155, Changchun, Jilin
  - Local Institution - 0181, Shenyang, Liaoning
  - Local Institution - 0182, Qingdao, Shandong
  - Local Institution - 0165, Shanghai, Shanghai Municipality
  - Local Institution - 0175, Shanghai, Shanghai Municipality
  - Local Institution - 0167, Ürümqi, Xinjiang
  - Local Institution - 0161, Hangzhou, Zhejiang
  - Local Institution - 0168, Hangzhou, Zhejiang
  - Local Institution - 0174, Hangzhou
  - Local Institution - 0172, Tianjin
- Colombia (3):
  - Local Institution - 0025, Bogota, Cundinamarca
  - Local Institution - 0022, Bogotá
  - Local Institution - 0024, Pasto
- Czechia (2):
  - Local Institution - 0200, Brno
  - Local Institution - 0197, Brno
- France (8):
  - Local Institution - 0077, Lille, Nord
  - Local Institution - 0080, Caen
  - Local Institution - 0081, Dijon
  - Local Institution - 0083, Montpellier
  - Local Institution - 0113, Nantes
  - Local Institution - 0079, Nice
  - Local Institution - 0078, Paris
  - Local Institution - 0119, Plérin
- Germany (9):
  - Local Institution - 0092, Mainz, Rhineland-Palatinate
  - Local Institution - 0094, Berlin
  - Local Institution - 0095, Cologne
  - Local Institution - 0089, Dresden
  - Local Institution - 0188, Düsseldorf
  - Local Institution - 0091, Essen
  - Local Institution - 0096, Freiburg im Breisgau
  - Local Institution - 0093, Hamburg
  - Local Institution - 0149, München
- Greece (4):
  - Local Institution - 0017, Nea Kifissia, Attikí
  - Local Institution - 0056, Athens
  - Local Institution - 0019, Ioannina
  - Local Institution - 0018, Pátrai
- Hong Kong (2):
  - Local Institution - 0191, Hong Kong
  - Local Institution - 0195, Hong Kong
- Hungary (3):
  - Local Institution - 0008, Budapest
  - Local Institution - 0007, Budapest
  - Local Institution - 0108, Debrecen
- Israel (5):
  - Local Institution - 0118, Haifa
  - Local Institution - 0116, Jerusalem
  - Local Institution - 0115, Petah Tikva
  - Local Institution - 0117, Ramat Gan
  - Local Institution - 0114, Tel Aviv
- Italy (6):
  - Local Institution - 0063, Pisa, Tuscany
  - Local Institution - 0062, Bergamo
  - Local Institution - 0205, Modena
  - Local Institution - 0061, Napoli
  - Local Institution - 0059, Roma
  - Local Institution - 0064, San Giovanni Rotondo
- Japan (10):
  - Local Institution - 0130, Nagoya, Aichi-ken
  - Local Institution - 0128, Chiba, Chiba
  - Local Institution - 0125, Kashiwa, Chiba
  - Local Institution - 0137, Sapporo, Hokkaido
  - Local Institution - 0127, Kita-Gun, Kagawa-ken
  - Local Institution - 0124, Suita-shi, Osaka
  - Local Institution - 0123, Kitaadachi-gun, Saitama
  - Local Institution - 0126, Chuo-ku, Tokyo
  - Local Institution - 0122, Minato-ku, Tokyo
  - Local Institution - 0129, Tokyo
- Mexico (3):
  - Local Institution - 0215, Mexico City, Mexico City
  - Local Institution - 0217, Toluca, State of Mexico
  - Local Institution - 0216, Querétaro
- Peru (4):
  - Local Institution - 0189, Lima
  - Local Institution - 0039, Lima
  - Local Institution - 0037, Lima
  - Local Institution - 0139, Lima
- Poland (3):
  - Local Institution - 0016, Lublin
  - Local Institution - 0013, Tarnobrzeg
  - Local Institution - 0014, Warsaw
- Portugal (2):
  - Local Institution - 0043, Lisbon
  - Local Institution - 0210, Porto
- Romania (5):
  - Local Institution - 0041, Craiova, Dolj
  - Local Institution - 0012, Baia Mare, Jud Maramures
  - Local Institution - 0040, Bucharest
  - Local Institution - 0042, Cluj-Napoca
  - Local Institution - 0055, Suceava
- Russia (5):
  - Local Institution - 0071, Chelyabinsk
  - Local Institution - 0086, Moscow
  - Local Institution - 0069, Moscow
  - Local Institution - 0105, Moscow
  - Local Institution - 0085, Saint Petersburg
- Singapore (2):
  - Local Institution - 0193, Singapore, Central Singapore
  - Local Institution - 0194, Singapore
- South Korea (2):
  - Local Institution - 0132, Seoul
  - Local Institution - 0131, Seoul
- Spain (6):
  - Local Institution - 0050, Badajoz
  - Local Institution - 0209, Badalona-barcelona
  - Local Institution - 0044, Barcelona
  - Local Institution - 0049, Pozuelo de Alarcon, Madrid
  - Local Institution - 0045, Valencia
  - Local Institution - 0212, Zaragoza
- Taiwan (3):
  - Local Institution - 0148, Tainan
  - Local Institution - 0133, Taipei
  - Local Institution - 0134, Taoyuan
- Turkey (Türkiye) (5):
  - Local Institution - 0203, Ankara
  - Local Institution - 0211, Ankara
  - Local Institution - 0201, Antalya
  - Local Institution - 0208, Diyarbakır
  - Local Institution - 0207, Edrine
- United Kingdom (5):
  - Local Institution - 0074, London, Greater London
  - Local Institution - 0073, Manchester, Greater Manchester
  - Local Institution - 0076, Nottingham, Nottinghamshire
  - Local Institution - 0075, Sutton, Surrey
  - Local Institution - 0072, Southampton

REFERENCES:
- [Derived] Lin D, Quan W, Garretson M, Chirikov V, Chen C, Singh P, Davis C, Sugarman R. Q-TWiST analysis of first-line nivolumab plus chemotherapy versus chemotherapy in patients with advanced gastric cancer, gastroesophageal junction cancer, or esophageal adenocarcinoma from CheckMate 649: 4-year follow-up results. Gastric Cancer. 2025 Sep;28(5):935-944. doi: 10.1007/s10120-025-01634-6. Epub 2025 Jul 9. PMID 40632415
- [Derived] Janjigian YY, Ajani JA, Moehler M, Shen L, Garrido M, Gallardo C, Wyrwicz L, Yamaguchi K, Cleary JM, Elimova E, Karamouzis M, Bruges R, Skoczylas T, Bragagnoli A, Liu T, Tehfe M, Zander T, Kowalyszyn R, Pazo-Cid R, Schenker M, Feeny K, Wang R, Lei M, Chen C, Nathani R, Shitara K. First-Line Nivolumab Plus Chemotherapy for Advanced Gastric, Gastroesophageal Junction, and Esophageal Adenocarcinoma: 3-Year Follow-Up of the Phase III CheckMate 649 Trial. J Clin Oncol. 2024 Jun 10;42(17):2012-2020. doi: 10.1200/JCO.23.01601. Epub 2024 Feb 21. PMID 38382001
- [Derived] Moehler M, Xiao H, Blum SI, Elimova E, Cella D, Shitara K, Ajani JA, Janjigian YY, Garrido M, Shen L, Yamaguchi K, Liu T, Schenker M, Kowalyszyn R, Bragagnoli AC, Bruges R, Montesarchio V, Pazo-Cid R, Hunter S, Davenport E, Wang J, Kondo K, Li M, Wyrwicz L. Health-Related Quality of Life With Nivolumab Plus Chemotherapy Versus Chemotherapy in Patients With Advanced Gastric/Gastroesophageal Junction Cancer or Esophageal Adenocarcinoma From CheckMate 649. J Clin Oncol. 2023 Dec 10;41(35):5388-5399. doi: 10.1200/JCO.23.00170. Epub 2023 Sep 15. PMID 37713657
- [Derived] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Wyrwicz L, Yamaguchi K, Skoczylas T, Bragagnoli AC, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. A plain language summary of the CheckMate 649 study: nivolumab in combination with chemotherapy compared to chemotherapy alone for untreated advanced or metastatic cancer of the stomach or esophagus. Future Oncol. 2023 Apr;19(11):739-752. doi: 10.2217/fon-2022-1149. Epub 2023 Mar 15. PMID 36919706
- [Derived] Liu T, Bai Y, Lin X, Li W, Wang J, Zhang X, Pan H, Bai C, Bai L, Cheng Y, Zhang J, Zhong H, Ba Y, Hu W, Xu R, Guo W, Qin S, Yang N, Lu J, Shitara K, Lei M, Li M, Bao N, Chen T, Shen L. First-line nivolumab plus chemotherapy vs chemotherapy in patients with advanced gastric, gastroesophageal junction and esophageal adenocarcinoma: CheckMate 649 Chinese subgroup analysis. Int J Cancer. 2023 Feb 15;152(4):749-760. doi: 10.1002/ijc.34296. Epub 2022 Oct 31. PMID 36121651
- [Derived] Janjigian YY, Shitara K, Moehler M, Garrido M, Salman P, Shen L, Wyrwicz L, Yamaguchi K, Skoczylas T, Campos Bragagnoli A, Liu T, Schenker M, Yanez P, Tehfe M, Kowalyszyn R, Karamouzis MV, Bruges R, Zander T, Pazo-Cid R, Hitre E, Feeney K, Cleary JM, Poulart V, Cullen D, Lei M, Xiao H, Kondo K, Li M, Ajani JA. First-line nivolumab plus chemotherapy versus chemotherapy alone for advanced gastric, gastro-oesophageal junction, and oesophageal adenocarcinoma (CheckMate 649): a randomised, open-label, phase 3 trial. Lancet. 2021 Jul 3;398(10294):27-40. doi: 10.1016/S0140-6736(21)00797-2. Epub 2021 Jun 5. PMID 34102137
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2031 Participants Randomized and 1991 Treated
Groups:
- Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX): Nivolumab + Xelox: Nivolumab 360 mg IV over 30 minutes on Day 1 of each treatment cycle, every 3 weeks + Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks
  Nivolumab + Folfox: Nivolumab 240 mg IV over 30 minutes on Day 1 of each treatment cycle, every 2 weeks + Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks
- Arm 2: Chemotherapy (XELOX or FOLFOX): Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. This chemotherapy group consists of the two comparison chemotherapy sub-groups. Arm 2a (792 participants) is the comparison group to Arm 1 and Arm 2b (404 participants) is the comparison group to Arm 3. Some participants were counted in both Arm 2a and Arm 2b.
- Arm 3: Nivolumab + Ipilimumab: 1 mg/kg nivolumab administered IV over 30 minutes followed by ipilimumab 3 mg/kg administered IV over 30 minutes on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1 to 4), followed by nivolumab 240 mg administered IV over 30 minutes on Day 1 of each treatment cycle every 2 weeks (Cycle 5 and beyond). Arm is closed to enrollment as of 05-June-2018.
Period: Pre-Treatment
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab
Started (= Randomized) | 789 | 833 | 409
Completed (= Moving to treatment period) | 782 | 806 | 403
Not Completed | 7 | 27 | 6
Not completed — Disease Progression | 0 | 1 | 0
Not completed — Adverse event unrelated to study drug | 0 | 2 | 1
Not completed — Participants request to discontinue study treatment | 0 | 2 | 0
Not completed — Participant withdrew consent | 2 | 20 | 3
Not completed — Participant no longer meets study criteria | 4 | 0 | 0
Not completed — Other reasons | 1 | 2 | 2
Period: Treatment
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab
Started (Treated) | 782 | 806 | 403
Completed (Continuing in the study) | 623 | 653 | 319
Not Completed | 159 | 153 | 84
Not completed — Death | 121 | 94 | 68
Not completed — Lost to Follow-up | 5 | 7 | 3
Not completed — Participant withdrew consent | 20 | 40 | 8
Not completed — Other reasons | 13 | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 789 | 833 | 409 | 2031
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (11.9) | 59.8 (12.1) | 59.4 (11.7) | 59.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 246 | 131 | 626
  Male | 540 | 587 | 278 | 1405
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 13 | 1 | 26
  Asian | 186 | 200 | 124 | 510
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 11 | 6 | 24
  White | 556 | 570 | 264 | 1390
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 28 | 39 | 14 | 81

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy With PD-L1 CPS ≥ 5
Description: Overall survival (OS), defined as the time from randomization to the time of death, in participants treated with Nivolumab plus Chemotherapy vs Chemotherapy with PD-L1 CPS (combined positive score) ≥ 5. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: From the date of randomization up to the date of death, up to approximately 17 months
Population: All randomized participants with PD-L1 CPS ≥ 5
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm 2a: Chemotherapy (XELOX or FOLFOX): Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. Comparison group to Arm 1.
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 473 | 482
Months | 14.39 [13.11 to 16.23] | 11.10 [10.02 to 12.09]
Statistical Analysis 1: Comparison: Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) vs Arm 2a: Chemotherapy (XELOX or FOLFOX); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.71, 98.4% CI 2-sided [0.59 to 0.86]

2. Primary Outcome: Progression Free Survival (PFS) in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy With PD-L1 CPS ≥ 5
Description: Progression Free Survival (PFS) is defined as the time from randomization to the date of the first documented PD or death due to any cause. PD is determined by blinded independent committee review (BICR) per RECIST1.1 criteria in participants treated with Nivolumab plus Chemotherapy vs Chemotherapy with PD-L1 CPS ≥ 5. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking in reference the smallest sum on study that also demonstrated an absolute increase of at least 5 mm. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: From randomization to the date of the first documented progressive disease (PD) per BICR or death due to any cause (up to approximately 10 months)
Population: All randomized participants with PD-L1 CPS ≥ 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 473 | 482
Months | 7.69 [7.03 to 9.17] | 6.05 [5.55 to 6.90]
Statistical Analysis 1: Comparison: Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) vs Arm 2a: Chemotherapy (XELOX or FOLFOX); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.68, 98% CI 2-sided [0.56 to 0.81]

3. Secondary Outcome: OS in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy
Description: Overall survival (OS), defined as the time from randomization to the time of death, in participants treated with Nivolumab plus Chemotherapy vs Chemotherapy with PD-L1 CPS ≥ 1, 10, and all randomized participants. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: From the date of randomization up to the date of death, up to approximately 17 months
Population: All randomized participants with available OS measurements in various subsets
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 697 | 727
Months
  All randomized participants | 13.73 [12.42 to 14.49] | 11.63 [10.94 to 12.52]
  Participants with PD-LI CPS ≥ 1: number analyzed (Participants) | 561 | 607
  Participants with PD-LI CPS ≥ 1 | 13.80 [12.42 to 14.82] | 11.37 [10.74 to 12.25]
  Participants with PD-L1 CPS ≥ 5: number analyzed (Participants) | 473 | 482
  Participants with PD-L1 CPS ≥ 5 | 14.39 [13.11 to 16.23] | 11.14 [10.05 to 12.12]
  Participants with PD-L1 CPS ≥ 10: number analyzed (Participants) | 316 | 355
  Participants with PD-L1 CPS ≥ 10 | 15.01 [13.63 to 16.66] | 10.94 [9.89 to 11.96]

4. Secondary Outcome: PFS in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy
Description: Progression free survival (PFS), defined as the time from randomization to the date of the first documented progressive disease (PD) or death due to any cause, in participants treated with Nivolumab plus Chemotherapy vs Chemotherapy by BICR per RECIST1.1 in participants with PD-L1 CPS ≥ 10, 1, or all randomized subjects. Progreessive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking in reference the smallest sum on study that also demonstrated an absolute increase of at least 5 mm. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: as for outcome 2
Population: All randomized participants with available PFS measurements in various subsets
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 614 | 598
Months
  All randomized participants | 7.75 [7.10 to 8.57] | 6.93 [6.67 to 7.16]
  Participants with PD-L1 CPS ≥ 1: number analyzed (Participants) | 506 | 510
  Participants with PD-L1 CPS ≥ 1 | 7.52 [7.03 to 8.51] | 6.93 [6.21 to 7.06]
  Participants with PD-L1 CPS ≥ 5: number analyzed (Participants) | 473 | 482
  Participants with PD-L1 CPS ≥ 5 | 8.31 [7.03 to 9.40] | 6.14 [5.55 to 6.93]
  Participants with PD-L1 CPS ≥ 10: number analyzed (Participants) | 285 | 307
  Participants with PD-L1 CPS ≥ 10 | 8.41 [7.00 to 9.79] | 5.82 [5.45 to 6.90]

5. Secondary Outcome: Objective Response Rate in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy
Description: Objective response rate (ORR) as assessed by BICR in participants with PD-L1 CPS ≥ 10, 5, 1, or all randomized participants. ORR is a percentage of participants determined by the number of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of measurable participants with target lesion at baseline. BOR is defined as the best response designation as determined by the BICR, recorded between the date of randomization and the date of objectively documented progression (per RECIST 1.1 as determined by the BICR) or the date of subsequent anti-cancer therapy, whichever occurs first. CR is defined as the disappearance of all target lesions. PR is define as at 30% decrease in the sum of diameters of target lesions. The 806 chemotherapy treated participants are split into two separate arms (Arm 2a and Arm 2b) to act as comparison groups to the other treatment arms.
Time Frame: From randomization to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (up to approximately 43 months)
Population: All randomized participants in various subsets as determined by PD-L1 CPS status
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Arm 2a: Chemotherapy (XELOX or FOLFOX): Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. This arm is a subgroup of the chemotherapy group that acts as a comparison group to Arm 1.
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 789 | 792
Percentage of Participants
  Participants with CPS ≥ 1: number analyzed (Participants) | 641 | 656
  Participants with CPS ≥ 1 | 48.8 [44.9 to 52.8] | 38.0 [34.2 to 41.8]
  Participants with CPS ≥ 5: number analyzed (Participants) | 473 | 482
  Participants with CPS ≥ 5 | 50.1 [45.5 to 54.7] | 38.2 [33.8 to 42.7]
  Participants with CPS ≥ 10: number analyzed (Participants) | 375 | 393
  Participants with CPS ≥ 10 | 48.8 [43.6 to 54.0] | 37.7 [32.9 to 42.7]
  All randomized participants | 46.9 [43.4 to 50.4] | 37.2 [33.9 to 40.7]

6. Secondary Outcome: Time to Symptom Deterioration (TTSD) in Participants Treated With Nivolumab Plus Chemotherapy vs Chemotherapy
Description: TTSD is defined as the the time from randomization until a clinically meaningful decline from baseline in Gastric Cancer Subscale (GaCS) score. A clinically meaningful deterioration is defined as a reduction of 8.2 points in the GaCS score. Subjects who do not deteriorate will be censored at the time of their last GACS assessment. Subjects without baseline GaCS assessment will be censored on the randomization date. Those with baseline GaCS, who do not have any GaCS assessments after randomization will be censored on the day after randomization.
Time Frame: From randomization until a clinically meaningful decline from baseline in GaCS score (approximately 10 months)
Population: All Treated participants with TTSD measurements
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1: Nivolumab + Chemotherapy (XELOX or FOLFOX) | Arm 2a: Chemotherapy (XELOX or FOLFOX)
Number analyzed (Participants) | 194 | 193
Months | NA [22.64 to NA] — Median and upper limits not reached because of insufficient number of events. | 21.03 [12.45 to NA] — Upper limits not reached because of insufficient number of events.

7. Secondary Outcome: OS in Participants Treated With Nivolumab Plus Ipilimumab vs Chemotherapy
Description: Overall survival (OS), defined as the time from randomization to the time of death, in participants treated with Nivolumab plus Ipilimumab vs Chemotherapy with PD-L1 CPS (combined positive score) ≥ 1, 5, 10, and all randomized participants. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: From the date of randomization up to the date of death, up to approximately 14 months
Population: All randomized participants with available measurements in various subsets as determined by PD-L1 CPS status
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm 2b: Chemotherapy (XELOX or FOLFOX): Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. Comparison group to Arm 3.
Arm/Group | Arm 2b: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab
Number analyzed (Participants) | 404 | 409
Months
  All randomized participants | 11.83 [10.97 to 12.71] | 11.73 [9.56 to 13.54]
  Participants with CPS ≥ 1: number analyzed (Participants) | 319 | 322
  Participants with CPS ≥ 1 | 11.47 [10.48 to 12.65] | 11.73 [9.49 to 13.54]
  Participants with CPS ≥ 5: number analyzed (Participants) | 239 | 234
  Participants with CPS ≥ 5 | 11.63 [10.05 to 12.71] | 11.24 [9.17 to 13.40]
  Participants with CPS ≥ 10: number analyzed (Participants) | 198 | 181
  Participants with CPS ≥ 10 | 11.33 [9.92 to 12.65] | 11.63 [9.26 to 13.54]

8. Secondary Outcome: PFS in Participants Treated With Nivolumab Plus Ipilimumab vs Chemotherapy
Description: Progression Free Survival (PFS) is defined as the time from randomization to the date of the first documented PD or death due to any cause. PD is determined by blinded independent committee review (BICR) per RECIST1.1 criteria in participants treated with Nivolumab plus Ipilumab vs Chemotherapy with PD-L1 CPS ≥ 10, 5, 1 or all randomized participants. Progressive disease (PD) is defined as at least a 20% increase in the sum of diameters of target lesions, taking in reference the smallest sum on study that also demonstrated an absolute increase of at least 5 mm. CPS is defined as the number of PD-L1 staining cells (tumor cells, lymphocytes, macrophages) divided by the total number of viable tumor cells, multiplied by 100.
Time Frame: From randomization to the date of the first documented progressive disease (PD) per BICR or death due to any cause (up to approximately 9 months)
Population: All randomized participants with available measurements in various subsets as determined by PD-L1 CPS status
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 2b: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab
Number analyzed (Participants) | 404 | 409
Months
  All randomized participants | 7.06 [6.87 to 8.21] | 2.83 [2.63 to 3.58]
  PD-L1 CPS ≥ 1: number analyzed (Participants) | 319 | 322
  PD-L1 CPS ≥ 1 | 6.93 [5.98 to 7.26] | 2.79 [2.60 to 3.91]
  PD-L1 CPS ≥ 5: number analyzed (Participants) | 239 | 234
  PD-L1 CPS ≥ 5 | 6.28 [5.59 to 7.06] | 2.83 [2.60 to 4.04]
  PD-L1 CPS ≥ 10: number analyzed (Participants) | 198 | 181
  PD-L1 CPS ≥ 10 | 6.28 [5.52 to 7.13] | 2.89 [2.63 to 4.24]

9. Secondary Outcome: Objective Response Rate in Participants Treated With Nivolumab Plus Ipilimumab vs Chemotherapy
Description: as for outcome 5
Time Frame: as for outcome 5
Population: All randomized participants in various subsets as determined by PD-L1 CPS status
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Arm 2b: Chemotherapy (XELOX or FOLFOX): Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. This arm is a subgroup of the chemotherapy group that acts as a comparison group to Arm 3.
Arm/Group | Arm 2b: Chemotherapy (XELOX or FOLFOX) | Arm 3: Nivolumab + Ipilimumab
Number analyzed (Participants) | 404 | 409
Percentage of Participants
  Participants with CPS ≥ 1: number analyzed (Participants) | 319 | 322
  Participants with CPS ≥ 1 | 37.3 [32.0 to 42.9] | 21.7 [17.4 to 26.6]
  Participants with CPS ≥ 5: number analyzed (Participants) | 239 | 234
  Participants with CPS ≥ 5 | 37.7 [31.5 to 44.1] | 23.1 [17.8 to 29.0]
  Participants with CPS ≥ 10: number analyzed (Participants) | 198 | 181
  Participants with CPS ≥ 10 | 35.9 [29.2 to 43.0] | 24.3 [18.3 to 31.2]
  All randomized participants | 34.9 [30.3 to 39.8] | 20.8 [17.0 to 25.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from date of randomization to study completion (up to approximately 5 years). Serious Adverse events and other adverse events were assessed from date of first dose to 100 days following date of last dose (up to approximately 5 years).
Description: All-Cause Mortality =all randomized participants AEs and NSAEs (Other Adverse Events) = all treated participants
Groups:
- Nivo + Chemo: Nivolumab + Xelox: Nivolumab 360 mg IV over 30 minutes on Day 1 of each treatment cycle, every 3 weeks + Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks
  Nivolumab + Folfox: Nivolumab 240 mg IV over 30 minutes on Day 1 of each treatment cycle, every 2 weeks + Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks
- Chemo: Chemotherapy (XELOX or FOLFOX): Xelox: Oxaliplatin 130 mg/m2 IV on Day 1 of each treatment cycle + capecitabine 1000 mg/m2 orally twice daily (ie, 1000 mg/m2 in the morning and 1000 mg/m2 in the evening) on Days 1 to 14 of each treatment cycle, every 3 weeks. Folfox: Oxaliplatin 85 mg/m2 + leucovorin 400 mg/m2 + fluorouracil 400 mg/m2 IV on Day 1 of each treatment cycle, and fluorouracil 1200 mg/m2 IV continuous infusion over 24 hours (or per local standard) daily on Days 1 and 2 of each treatment cycle, every 2 weeks. This chemotherapy group consists of the two comparison chemotherapy sub-groups. Arm 2a (792 participants) is the comparison group to Arm 1 and Arm 2b (404 participants) is the comparison group to Arm 3. Some participants were counted in both Arm 2a and Arm 2b.
- Nivo + Ipi: 1 mg/kg nivolumab administered IV over 30 minutes followed by ipilimumab 3 mg/kg administered IV over 30 minutes on Day 1 of each treatment cycle every 3 weeks for 4 doses (Cycles 1 to 4), followed by nivolumab 240 mg administered IV over 30 minutes on Day 1 of each treatment cycle every 2 weeks (Cycle 5 and beyond). Arm is closed to enrollment as of 05-June-2018.
Arm/Group | Nivo + Chemo | Chemo | Nivo + Ipi
All-Cause Mortality (participants affected / at risk) | 691/782 | 741/806 | 361/403
Serious Adverse Events (participants affected / at risk) | 529/782 | 474/806 | 307/403
Other Adverse Events (participants affected / at risk) | 763/782 | 756/806 | 369/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivo + Chemo (N=782) | Chemo (N=806) | Nivo + Ipi (N=403)
Anaemia (Blood and lymphatic system disorders) | 28 | 17 | 13
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 10 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 4 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 3 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Autoimmune myocarditis (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 5 | 3
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 3 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Choledochal cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Microvillous inclusion disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 3 | 1 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 1 | 4
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0 | 4
Hypopituitarism (Endocrine disorders) | 3 | 0 | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Immune-mediated hypophysitis (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Ocular vasculitis (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 13 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Ascites (Gastrointestinal disorders) | 15 | 9 | 6
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0 | 3
Colitis (Gastrointestinal disorders) | 6 | 0 | 11
Constipation (Gastrointestinal disorders) | 3 | 3 | 2
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 14 | 13
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 13 | 23 | 9
Enteritis (Gastrointestinal disorders) | 1 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 4 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 3 | 11 | 4
Gastric perforation (Gastrointestinal disorders) | 1 | 3 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 9 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 4 | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 2 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1 | 11
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 6 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 2 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 1
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 10 | 7
Obstruction gastric (Gastrointestinal disorders) | 2 | 5 | 5
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Oesophageal compression (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 4 | 3 | 4
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 3 | 0 | 2
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Prepyloric stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 5 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 | 10 | 13
Vomiting (Gastrointestinal disorders) | 29 | 24 | 12
Asthenia (General disorders) | 1 | 5 | 3
Catheter site extravasation (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Complication associated with device (General disorders) | 1 | 2 | 1
Death (General disorders) | 1 | 1 | 2
Disease progression (General disorders) | 1 | 4 | 0
Effusion (General disorders) | 1 | 0 | 0
Euthanasia (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 6
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 5 | 7 | 3
Generalised oedema (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 3 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1
Pain (General disorders) | 3 | 4 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 22 | 11 | 9
Sudden death (General disorders) | 2 | 3 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 6
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 3 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 2 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 5
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2 | 5
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 5
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 | 0 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 6 | 3 | 2
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 2 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 3
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 4 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 2 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Amoebic colitis (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 4 | 1 | 3
Biliary tract infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 3 | 2
Chorioretinitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 2 | 2 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Encephalitis (Infections and infestations) | 2 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Lung abscess (Infections and infestations) | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1 | 1
Peritonitis bacterial (Infections and infestations) | 3 | 1 | 0
Pneumonia (Infections and infestations) | 30 | 21 | 13
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 13 | 8 | 3
Septic shock (Infections and infestations) | 1 | 2 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 2
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 6
Urosepsis (Infections and infestations) | 1 | 0 | 1
Vascular device infection (Infections and infestations) | 3 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 11 | 6 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 6 | 1 | 2
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 2
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 2 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Hepatitis C virus test positive (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 3 | 3 | 0
Platelet count decreased (Investigations) | 3 | 4 | 1
Transaminases increased (Investigations) | 0 | 0 | 2
Troponin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 9 | 6
Dehydration (Metabolism and nutrition disorders) | 8 | 7 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 246 | 242 | 112
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 2
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Immune-mediated neuropathy (Nervous system disorders) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 9 | 4 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0
Device breakage (Product Issues) | 0 | 1 | 0
Device dislocation (Product Issues) | 3 | 2 | 2
Device leakage (Product Issues) | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 0 | 1
Device occlusion (Product Issues) | 3 | 0 | 0
Stent malfunction (Product Issues) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Eating disorder (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 3 | 9
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 1
Nephritis (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 3 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 6
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 | 1 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 9
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 3 | 3
Embolism (Vascular disorders) | 6 | 1 | 0
Hypotension (Vascular disorders) | 2 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 1 | 0
Obstructive shock (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 28 | 17 | 13
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 10 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 4 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 4 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Autoimmune myocarditis (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 5 | 3
Myocardial injury (Cardiac disorders) | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 3 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Microvillous inclusion disease (Congenital, familial and genetic disorders) | 0 | 0 | 1
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 3 | 1 | 4
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0 | 4
Hypopituitarism (Endocrine disorders) | 3 | 0 | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1
Immune-mediated hypophysitis (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Ocular vasculitis (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 13 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Ascites (Gastrointestinal disorders) | 15 | 9 | 6
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0 | 3
Colitis (Gastrointestinal disorders) | 6 | 0 | 11
Constipation (Gastrointestinal disorders) | 3 | 3 | 2
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 21 | 14 | 13
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 13 | 23 | 9
Enteritis (Gastrointestinal disorders) | 1 | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 4 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 3 | 11 | 4
Gastric perforation (Gastrointestinal disorders) | 1 | 3 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 9 | 4
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 4 | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 2 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1 | 11
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 7 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 2 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 1
Malignant ascites (Gastrointestinal disorders) | 1 | 1 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 10 | 7
Obstruction gastric (Gastrointestinal disorders) | 4 | 6 | 6
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Oesophageal compression (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 4 | 3 | 4
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 3 | 0 | 2
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1 | 0
Prepyloric stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 5 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 17 | 10 | 13
Vomiting (Gastrointestinal disorders) | 29 | 23 | 11
Asthenia (General disorders) | 1 | 5 | 3
Catheter site extravasation (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Complication associated with device (General disorders) | 1 | 2 | 1
Death (General disorders) | 1 | 1 | 2
Disease progression (General disorders) | 0 | 1 | 0
Effusion (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 2 | 6
Gait disturbance (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 5 | 7 | 3
Generalised oedema (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 3 | 1
Mucosal inflammation (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 3 | 0 | 1
Pain (General disorders) | 3 | 4 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 22 | 11 | 9
Sudden death (General disorders) | 2 | 3 | 2
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 6
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 3 | 0 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 2 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 3
Hepatic cyst ruptured (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2 | 5
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 5
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 2
Immune-mediated hepatic disorder (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 3 | 0 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 6 | 4 | 2
Liver disorder (Hepatobiliary disorders) | 2 | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 3
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 4 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 2 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0
Amoebic colitis (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 4 | 1 | 3
Biliary tract infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 3 | 2
Chorioretinitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 2 | 2 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Encephalitis (Infections and infestations) | 2 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Giardiasis (Infections and infestations) | 0 | 0 | 1
Haematological infection (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Lung abscess (Infections and infestations) | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 1 | 1
Peritonitis bacterial (Infections and infestations) | 2 | 1 | 0
Pneumonia (Infections and infestations) | 30 | 21 | 14
Pneumonia aspiration (Infections and infestations) | 3 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 12 | 8 | 3
Septic shock (Infections and infestations) | 1 | 2 | 2
Sialoadenitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 2
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 6
Urosepsis (Infections and infestations) | 1 | 0 | 1
Vascular device infection (Infections and infestations) | 3 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Afferent loop syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 11 | 6 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 6 | 1 | 2
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 2
Electrocardiogram ST segment elevation (Investigations) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 2 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Hepatitis C virus test positive (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 3 | 3 | 0
Platelet count decreased (Investigations) | 3 | 4 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 9 | 6
Dehydration (Metabolism and nutrition disorders) | 8 | 7 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 3
Hypophagia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 248 | 246 | 112
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 2
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 2 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 2
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Immune-mediated neuropathy (Nervous system disorders) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Neuritis (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 9 | 4 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 2 | 0
Device breakage (Product Issues) | 0 | 1 | 0
Device dislocation (Product Issues) | 3 | 2 | 2
Device leakage (Product Issues) | 0 | 1 | 0
Device occlusion (Product Issues) | 3 | 0 | 0
Stent malfunction (Product Issues) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Eating disorder (Psychiatric disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 4 | 9
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 1
Nephritis (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 3 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Mediastinal effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 | 1 | 7
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 10
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Euthanasia (Surgical and medical procedures) | 0 | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3 | 3
Embolism (Vascular disorders) | 6 | 1 | 0
Hypotension (Vascular disorders) | 2 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 1 | 0
Obstructive shock (Vascular disorders) | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivo + Chemo (N=782) | Chemo (N=806) | Nivo + Ipi (N=403)
Anaemia (Blood and lymphatic system disorders) | 312 | 276 | 132
Leukopenia (Blood and lymphatic system disorders) | 75 | 64 | 9
Neutropenia (Blood and lymphatic system disorders) | 218 | 203 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 173 | 160 | 10
Hyperthyroidism (Endocrine disorders) | 30 | 2 | 26
Hypothyroidism (Endocrine disorders) | 82 | 13 | 54
Abdominal distension (Gastrointestinal disorders) | 56 | 43 | 26
Abdominal pain (Gastrointestinal disorders) | 159 | 134 | 66
Abdominal pain upper (Gastrointestinal disorders) | 73 | 75 | 36
Constipation (Gastrointestinal disorders) | 201 | 177 | 77
Diarrhoea (Gastrointestinal disorders) | 309 | 286 | 111
Dysphagia (Gastrointestinal disorders) | 64 | 64 | 32
Nausea (Gastrointestinal disorders) | 385 | 362 | 101
Stomatitis (Gastrointestinal disorders) | 67 | 57 | 13
Vomiting (Gastrointestinal disorders) | 247 | 233 | 72
Asthenia (General disorders) | 119 | 127 | 47
Fatigue (General disorders) | 271 | 234 | 103
Malaise (General disorders) | 40 | 41 | 19
Mucosal inflammation (General disorders) | 78 | 47 | 7
Oedema peripheral (General disorders) | 93 | 66 | 44
Pyrexia (General disorders) | 143 | 93 | 93
Hypersensitivity (Immune system disorders) | 51 | 12 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 67 | 31 | 12
Alanine aminotransferase increased (Investigations) | 118 | 86 | 76
Amylase increased (Investigations) | 91 | 45 | 48
Aspartate aminotransferase increased (Investigations) | 163 | 113 | 81
Blood alkaline phosphatase increased (Investigations) | 107 | 66 | 47
Blood bilirubin increased (Investigations) | 83 | 61 | 30
Blood creatinine increased (Investigations) | 42 | 22 | 35
Lipase increased (Investigations) | 108 | 72 | 52
Neutrophil count decreased (Investigations) | 171 | 139 | 19
Platelet count decreased (Investigations) | 172 | 132 | 21
Weight decreased (Investigations) | 139 | 128 | 60
White blood cell count decreased (Investigations) | 123 | 92 | 16
Decreased appetite (Metabolism and nutrition disorders) | 236 | 226 | 111
Hyperglycaemia (Metabolism and nutrition disorders) | 84 | 63 | 37
Hypoalbuminaemia (Metabolism and nutrition disorders) | 109 | 72 | 62
Hypocalcaemia (Metabolism and nutrition disorders) | 53 | 37 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 93 | 74 | 37
Hyponatraemia (Metabolism and nutrition disorders) | 72 | 51 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 | 42 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 86 | 66 | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 20 | 9
Dizziness (Nervous system disorders) | 56 | 58 | 16
Dysgeusia (Nervous system disorders) | 48 | 43 | 10
Headache (Nervous system disorders) | 89 | 52 | 33
Hypoaesthesia (Nervous system disorders) | 45 | 42 | 6
Neuropathy peripheral (Nervous system disorders) | 238 | 210 | 7
Paraesthesia (Nervous system disorders) | 72 | 78 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 146 | 128 | 13
Insomnia (Psychiatric disorders) | 61 | 69 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 63 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 66 | 49 | 37
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 108 | 96 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 79 | 18 | 72
Rash (Skin and subcutaneous tissue disorders) | 91 | 23 | 77
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 7 | 41
Hypertension (Vascular disorders) | 48 | 41 | 17
Hypotension (Vascular disorders) | 26 | 21 | 21
Anaemia (Blood and lymphatic system disorders) | 312 | 279 | 132
Leukopenia (Blood and lymphatic system disorders) | 76 | 65 | 9
Neutropenia (Blood and lymphatic system disorders) | 221 | 205 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 172 | 161 | 10
Hyperthyroidism (Endocrine disorders) | 30 | 2 | 26
Hypothyroidism (Endocrine disorders) | 82 | 13 | 54
Abdominal distension (Gastrointestinal disorders) | 56 | 43 | 26
Abdominal pain (Gastrointestinal disorders) | 159 | 134 | 66
Abdominal pain upper (Gastrointestinal disorders) | 75 | 77 | 37
Constipation (Gastrointestinal disorders) | 201 | 177 | 77
Diarrhoea (Gastrointestinal disorders) | 310 | 287 | 112
Dysphagia (Gastrointestinal disorders) | 64 | 65 | 32
Nausea (Gastrointestinal disorders) | 386 | 364 | 101
Stomatitis (Gastrointestinal disorders) | 68 | 57 | 13
Vomiting (Gastrointestinal disorders) | 248 | 234 | 72
Asthenia (General disorders) | 119 | 130 | 48
Fatigue (General disorders) | 273 | 235 | 103
Malaise (General disorders) | 40 | 41 | 19
Mucosal inflammation (General disorders) | 77 | 47 | 7
Oedema peripheral (General disorders) | 93 | 67 | 44
Pyrexia (General disorders) | 143 | 95 | 93
Hypersensitivity (Immune system disorders) | 48 | 13 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 67 | 31 | 12
Alanine aminotransferase increased (Investigations) | 120 | 88 | 76
Amylase increased (Investigations) | 91 | 45 | 48
Aspartate aminotransferase increased (Investigations) | 165 | 115 | 81
Blood alkaline phosphatase increased (Investigations) | 107 | 69 | 47
Blood bilirubin increased (Investigations) | 83 | 62 | 30
Blood creatinine increased (Investigations) | 42 | 22 | 35
Lipase increased (Investigations) | 107 | 72 | 52
Neutrophil count decreased (Investigations) | 171 | 140 | 19
Platelet count decreased (Investigations) | 175 | 132 | 21
Weight decreased (Investigations) | 139 | 128 | 60
White blood cell count decreased (Investigations) | 124 | 92 | 16
Decreased appetite (Metabolism and nutrition disorders) | 237 | 226 | 111
Hyperglycaemia (Metabolism and nutrition disorders) | 82 | 64 | 37
Hypoalbuminaemia (Metabolism and nutrition disorders) | 109 | 72 | 62
Hypocalcaemia (Metabolism and nutrition disorders) | 53 | 37 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 93 | 74 | 37
Hyponatraemia (Metabolism and nutrition disorders) | 72 | 51 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 74 | 42 | 30
Back pain (Musculoskeletal and connective tissue disorders) | 87 | 69 | 38
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 21 | 9
Dizziness (Nervous system disorders) | 57 | 59 | 16
Dysgeusia (Nervous system disorders) | 48 | 43 | 10
Headache (Nervous system disorders) | 89 | 53 | 33
Hypoaesthesia (Nervous system disorders) | 45 | 42 | 6
Neuropathy peripheral (Nervous system disorders) | 241 | 211 | 7
Paraesthesia (Nervous system disorders) | 72 | 78 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 146 | 129 | 13
Insomnia (Psychiatric disorders) | 61 | 69 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 102 | 64 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 66 | 49 | 37
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 108 | 98 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 79 | 19 | 72
Rash (Skin and subcutaneous tissue disorders) | 90 | 22 | 77
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 7 | 41
Hypertension (Vascular disorders) | 48 | 42 | 17
Hypotension (Vascular disorders) | 26 | 21 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT02872116/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02872116/SAP_001.pdf